CLINICAL TRIAL: NCT03998098
Title: A Single-Center Study To Demonstrate the Safety and Performance of Lifelight® First Software Application - A Non-invasive Vital Signs Monitoring Device
Brief Title: A Single Center Study to Demonstrate the Safety and Performance of Lifelight® First Software Application
Status: Completed | Type: Observational
Sponsor: Xim Limited (Industry)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: X4
Record Dates: First submitted 2019-05-13; First posted 2019-06-25 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Vital Signs
Keywords: Blood Pressure; SPO2; Oxygen Saturation; Respiratory Rate; Pulse; Breathing Rate; Heart Rate
MeSH Terms: interventions — Oxygen Saturation; Oximetry; Heart Rate; Pulse; Respiratory Rate; Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Oxygen Saturation (Oximetry): Arm to determine the performance of the Oxygen Saturation measurement in LifeLight First
  Interventions: Diagnostic Test: Oxygen Saturation (Oximetry)
- Heart Rate (Pulse): Arm to determine the performance of the Heart Rate measurement in LifeLight First
  Interventions: Diagnostic Test: Heart Rate (Pulse)
- Respiratory Rate: Arm to determine the performance of the Respiratory Rate measurement in LifeLight First
  Interventions: Diagnostic Test: Respiratory Rate
- Blood Pressure: Arm to determine the performance of the Blood Pressure measurement in LifeLight First
  Interventions: Diagnostic Test: Blood Pressure

INTERVENTIONS:
Diagnostic Test: Oxygen Saturation (Oximetry) — Participants enter a chamber with a modifiable atmosphere and sit on a bench associated with an exercise bicycle. The subject breathes hypoxic air to achieve various SpO2 readings throughout the range of 80-97%.
  The participants undertake recumbent cycling for up to 10 minutes at various intervals and differing oxygen/nitrogen balances to induce changes in their vital signs.
  Measurements of the Vital Signs are taken at various time points using Lifelight First and the reference device using 2 observers
  Other Names: Welch Allyn Connex Spot Monitor CSM 7500; LifeLight First
  Groups: Oxygen Saturation (Oximetry)
Diagnostic Test: Heart Rate (Pulse) — Participants enter a chamber with a modifiable atmosphere and sit on a bench associated with an exercise bicycle. The subject breathes hypoxic air to achieve various SpO2 readings throughout the range of 80-97%.
  The participants undertake recumbent cycling for up to 10 minutes at various intervals and differing oxygen/nitrogen balances to induce changes in their vital signs.
  Measurements of the Vital Signs are taken at various time points using Lifelight First and the reference device using 2 observers
  Other Names: Welch Allyn Connex Spot Monitor CSM 7500; LifeLight First
  Groups: Heart Rate (Pulse)
Diagnostic Test: Respiratory Rate — Participants enter a chamber with a modifiable atmosphere and sit on a bench associated with an exercise bicycle. The subject breathes hypoxic air to achieve various SpO2 readings throughout the range of 80-97%.
  The participants undertake recumbent cycling for up to 10 minutes at various intervals and differing oxygen/nitrogen balances to induce changes in their vital signs.
  Measurements of the Vital Signs are taken at various time points using Lifelight First and the reference device using 2 observers
  Other Names: Two Clinical Observers; LifeLight First
  Groups: Respiratory Rate
Diagnostic Test: Blood Pressure — Participants enter a chamber with a modifiable atmosphere and sit on a bench associated with an exercise bicycle. The subject breathes hypoxic air to achieve various SpO2 readings throughout the range of 80-97%.
  The participants undertake recumbent cycling for up to 10 minutes at various intervals and differing oxygen/nitrogen balances to induce changes in their vital signs.
  Measurements of the Vital Signs are taken at various time points using Lifelight First and the reference device using 2 observers For participants only participating in the Blood Pressure Arm of the trial, they will not be required to enter the normobaric chamber but will have their blood pressure readings taken in the ambient environment including lying supine in order to generate hypotensive readings.
  Other Names: Welch Allyn Connex Spot Monitor CSM 7500; LifeLight First
  Groups: Blood Pressure

SUMMARY:
This study validates Lifelight® First, a software application, in a laboratory setting. Participants will undergo testing to obtain measurements from one or more of the four vital signs.

DETAILED DESCRIPTION:
Assessment of vital signs is an essential part of any clinical assessment and is undertaken regularly on patients accessing healthcare services. The accuracy of these measurements is of vital importance as decisions regarding the urgency of medical review and subsequent management are often influenced by these measures.

The measurement of vital signs as part of normal medical care requires a level of medical / nursing skill or patient training. Observations can be altered by stress or anxiety making the results less representative of the patient's clinical state. This is particularly recognised in the measurement of blood pressure but stress can also alter heart and respiratory rate.

Regular community and/or home monitoring of vital signs is useful in older populations and those with long-term conditions; standard of care methods can be labour intensive for health care providers, leading to greater financial burdens for health services.

Lifelight® First is software which allows non-invasive, non-contact measurement of these observations. It can be used on a tablet (e.g. Apple® iPad®) that possesses an integral camera. The use of computer technology is now commonplace in society so the general public are likely to be accepting of this as a non-threatening method of measurement, thus reducing the impact of anxiety on the results. Lifelight® First therefore has potential application within various areas of the health care system, it could also be useful in settings where direct access to health care is limited or as a part of a telemedicine service.

This study has been designed to evaluate the safety and performance of Lifelight® First, an investigational medical device. The data will be used to support the CE marking of the Lifelight® First device. The study design has been based upon the guidance in ISO standards and also within published scientific literature. Ultimately the data points to be obtained and methodology will be required to follow this guidance in order to obtain the CE mark.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is informed and has been given ample time and opportunity to think about his/her participation and has given his/her written informed consent
2. Subject is ≥18 years of age
3. Subject's health status: individual is considered to be healthy (hypertension and hypotension is permissible. Other stable diseases at the time of testing are also permissible)
4. Subject is capable of undergoing controlled hypoxaemia to the levels called for the in the protocol with minimal medical risk (unless only participating in the blood pressure study).

Exclusion Criteria:

1. Subject cannot expose their face fully for a reading to be taken
2. Subject is unable to give informed consent
3. Subject is outside of the specified age range
4. Subject has already taken part in the study (all 4 sub studies)
5. Subject with significant irregular heart rhythm or any disease that might affect the results of the study
6. Subject is not capable of undergoing controlled hypoxia and would be placed at undue medical risk if this occurred
7. Subject has any contraindications identified that would deem them unsuitable to take part

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusion/exclusion criteria is limited to the intended use of the device, therefore only individuals, of any sex, over the age of 18 will be included in the study. The individuals for the purpose of the study have to be able to perform physical activity in the form of the ergometer if they are undertaking the exercise component.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Readings Validation | Single Visit; up to one day
  Agreement of Lifelight® First standard of care and range for blood pressure as per ISO 81060-2-Non-invasive-sphygmomanometers-Part 2-Clinical validation of automated measurement type
Oxygen Saturation Readings Validation | Single Visit; up to one day
  Agreement of Lifelight® First standard of care and range for oxygen saturation as per ISO 80601-2-61-Medical electrical equipment-Part 2-61:Particular requirements for basic safety and essential performance of pulse oximeter equipment
Heart Rate (pulse) Readings Validation | Single Visit; up to one day
  Agreement of Lifelight® First standard of care and range for heart rate (pulse) function as per ISO 80601-2-61- Particular requirements for basic safety and essential performance of pulse oximeter equipment
Respiratory Rate Readings Validation | Single Visit; up to one day
  Agreement of Lifelight® First standard of care and range for respiratory rate by manually counting chest rises.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth, Department of Sport and Exercise Science, Portsmouth, England, United Kingdom